CLINICAL TRIAL: NCT00197444
Title: A Phase II Study of Daily Low-Dose of Nedaplatin (CDGP:Cis-Diammine-Glycolatoplatinum) and Continuous Infusion of 5-FU Combined With Radiation for the Treatment of Esophageal Cancer
Brief Title: Low-Dose Nedaplatin (CDGP:Cis-Diammine-Glycolatoplatinum)/5-FU Combined With Radiation for Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamamatsu University (Other)
Responsible Party: Satoshi Osawa, M.D./Ph.D., First Department of Medicine, Hamamatsu University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAMA-M1-C001
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Esophageal Cancer; Squamous Cell Carcinoma
Keywords: esophageal cancer; Nedaplatin; 5-FU; chemotherapy; radiation; chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell | interventions — Radiation; nedaplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Chemoradiotherapy
  Interventions: Drug: CDGP/5-FU combined with radiation; Radiation: Radiotherapy

INTERVENTIONS:
Drug: CDGP/5-FU combined with radiation — Low-dose of Nedaplatin (CDGP) 10 mg/body/day was daily administered on day 1-5, 8-13, 15-19, 22-26 and 5-FU 500 mg/body/day was continuously administered on day 1-5, 8-13, 15-19, 22-26.
  Other Names: Nedaplatin; 5-FU
Radiation: Radiotherapy — Fractionated external radiotherapy was performed from the first day of chemotherapy and a total dose of 50.4-66 Gy was delivered at the rate of 1.8-2.0 Gy per fraction.
  Other Names: Radiation

SUMMARY:
The purpose of this study is to clarify efficacy and toxicity of daily low-dose Nedaplatin (CDGP) and continuous infusion of 5-FU combined with radiation in patients with esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
The tumor stages and disease grades were classified according to the TNM classification (sixth edition) of the International Union against Cancer (UICC). These were determined conventionally by computed tomography (CT) of the neck, chest and abdomen, bone scan, endoscopic ultrasonography (EUS), endoscopy and esophagography.

Low-dose of Nedaplatin (CDGP) 10 mg/body/day was daily administered on day 1-5, 8-13, 15-19, 22-26 and 5-FU 500 mg/body/day was continuously administered on day 1-5, 8-13, 15-19, 22-26. Fractionated radiotherapy was performed from day 1 and a total dose of 50-60 Gy was delivered at the rate of 1.8-2.0 Gy per fraction. Serotonin receptor antagonist was preventively given as an antinauseant just before the administration of Nedaplatin.

Tumor response was assessed according to the Response Evaluation Criteria In Solid Tumors (UICC, 2002). Toxicities were graded according to the Common Terminology Criteria for Adverse Events v3.0 (CTCAE). Survival was calculated from the start of chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed cases histologically as squamous cell carcinoma,
* a performance status 0 to 2,
* white blood cells >3,000/microL,
* platelets >100,000/microL,
* serum total bilirubin <2.0 mg/dl,
* serum transaminase <3 times the upper normal limit,
* serum creatinine <1.5 mg/dl,
* creatinine clearance >60 ml/min

Exclusion Criteria:

* serious cardiac disease
* prior chemotherapy and radiotherapy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-01; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 3 months

SECONDARY OUTCOMES:
Adverse events | every 3-6 months
Survival rate | every 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Osawa, M.D., Principal Investigator — First Department of Medicine, Hamamatsu University School of Medicine
Locations (1):
- First Department of Medicine, Hamamatsu University School of Medicine, Hamamatsu, Japan

REFERENCES:
- [Derived] Osawa S, Furuta T, Sugimoto K, Kosugi T, Terai T, Yamade M, Takayanagi Y, Nishino M, Hamaya Y, Kodaira C, Yamada T, Iwaizumi M, Takagaki K, Yoshida K, Kanaoka S, Ikuma M. Prospective study of daily low-dose nedaplatin and continuous 5-fluorouracil infusion combined with radiation for the treatment of esophageal squamous cell carcinoma. BMC Cancer. 2009 Nov 22;9:408. doi: 10.1186/1471-2407-9-408. PMID 19930599